CLINICAL TRIAL: NCT01813760
Title: Treatment of Periorbital and Perioral Wrinkles With the Applications of the Iluminage Diode Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN12-AFF-UL-09
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Peri-orbital Wrinkles; Peri-oral Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diode laser (Experimental): Diode laser to treat peri-orbital and peri-oral wrinkles
  Interventions: Device: Illuiminage ® Diode Laser

INTERVENTIONS:
Device: Illuiminage ® Diode Laser — Diode laser for treatment of peri-orbital and peri-oral wrinkles

SUMMARY:
The Diode laser system is being used in this marketing study for the treatment of wrinkles around the eyes and mouth.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are healthy females between 35 and 60 years of age.
2. Subjects who have Fitzpatrick skin type I-VI
3. Subjects who have provided written and verbal informed consent
4. Subjects who are willing and able to comply with study instructions and to return to the clinic for required visits and have photographs of their face taken
5. Subjects who have perioral and periorbital wrinkles, as deemed appropriate by the Investigator or his designees

Exclusion Criteria:

1. Subjects who currently use or have used in the prior 30 days any skin products that contain alpha hydroxy acids (AHA) e.g. glycolic, lactic, citric, or mendelic acid containing products or retinol/tretinoin containing products or exfoliating washes, masks or scrubs or other micro-dermabrasion skin care products. on the laser application areas
2. Subjects who are unwilling to maintain their daily skin care regimen for the duration of the study,
3. Subjects who have any skin pathology or condition that could interfere with the evaluation i.e. personal or family history of skin cancer, rosacea and/or requires the use of interfering topical or systemic therapies.
4. Subjects with synthetic or metal implants or permanent cosmetic tattoos in the test areas
5. Subjects who have a history of abnormal scarring, e.g. keloids or have significant scarring in the areas to be treated
6. Subjects with bleeding disorders or taking anticoagulation medications, including heavy use of aspirin
7. Subjects who have participated in any clinical investigation involving the face within the 30 days prior to the first planned laser application or subjects who plan to participate in concomitant facial studies during this trial
8. Subjects, who are pregnant, were pregnant or gave birth in the last 3 months, are currently breast feeding, or might become pregnant during the course of the study
9. Subjects who have a history of light triggered seizures
10. Subjects with prior use of neurotoxins e.g. Botox®, collagen, fat injections and/or other methods of skin augmentation (enhancement with injected or implanted material) of the face or having had chemical peels within 6 months of initial laser application or planning to so during the course of the study
11. Subject's use of oral isotretinoin (Accutane®) within 12 months of initial laser application or during the course of the study
12. Subjects having had facial skin treatments with any professional laser, light based, radiofrequency or other devices within the last year
13. Subjects ever having facial skin treatments with home use laser, light based or radiofrequency or other devices, i.e. PaloVia® or Tria®

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Photographic Evaluation | 60 days post first treatment
  Compare severity of wrinkles from baseline to 60 days post treatment based on Fitpatrick Scale.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | up to 4 months post 1st treatment
  Adverse events and side effects will be recorded
Photographic Evaluation | Up to 40 days
  Compare severity of wrinkles from baseline to 1,10, 20 and 40 days post treatment based on Fitzpatrick Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Cynosure, Inc, Westford, Massachusetts, United States